CLINICAL TRIAL: NCT07275697
Title: Waiting on Atrial Fibrillation Intervention Therapy (WAIT) Study
Acronym: WAIT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emma Svennberg (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Emma Svennberg, Associate professor, Consultant, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WAIT; 2025-524182-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); Obesity & Overweight
Keywords: Semaglutide; Implantable Loop Recorder; Ablation; Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Overweight | interventions — semaglutide; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Randomized to Semaglutide (Experimental): Participants randomized to the active arm receive once-weekly subcutaneous semaglutide (Wegovy®) initiated at 0.25 mg and uptitrated to a target dose of 2.4 mg as tolerated, according to the approved SmPC. Treatment begins ≥3 months before the planned first catheter ablation for atrial fibrillation. Participants receive structured lifestyle and weight-management advice in accordance with routine clinical practice.
  Interventions: Drug: Semaglutide 2.4 mg; Behavioral: Standard medical treatment
- Standard of care (Active Comparator): Participants randomized to the standard-of-care arm receive routine clinical management for atrial fibrillation and weight-related comorbidities without GLP-1 receptor agonist therapy. Usual care may include lifestyle counselling, blood pressure and lipid management, treatment of dysglycaemia, and guideline-directed preparation for first-time catheter ablation. No trial-specific medicinal product is administered. Pa
  Interventions: Behavioral: Standard medical treatment

INTERVENTIONS:
Drug: Semaglutide 2.4 mg — The intervention consists of once-weekly subcutaneous semaglutide (Wegovy®), initiated at 0.25 mg and uptitrated to a target dose of 2.4 mg as tolerated, administered for at least three months prior to the participant's first planned atrial fibrillation ablation. Semaglutide is provided in pre-filled pens and used according to the approved SmPC for weight management. This intervention is uniquely characterized by pharmacological weight-loss therapy added on top of standard-of-care management, distinguishing it from the control arm, which receives identical clinical follow-up and lifestyle counselling but no GLP-1 receptor agonist. This allows evaluation of whether targeted metabolic therapy before ablation improves arrhythmia-related outcomes.
  Other Names: Standard of care
  Arms: Randomized to Semaglutide
Behavioral: Standard medical treatment — Participants randomized to the standard-of-care arm receive routine clinical management for atrial fibrillation and weight-related comorbidities without GLP-1 receptor agonist therapy. Usual care may include lifestyle counselling, blood pressure and lipid management, treatment of dysglycaemia, and guideline-directed preparation for first-time catheter ablation. No trial-specific medicinal product is administered.

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disorder and is associated with symptoms, reduced quality of life, heart failure, stroke, and a high risk of recurrence after catheter ablation. Many patients scheduled for their first ablation are overweight or have obesity, which is one of the strongest predictors of AF recurrence. Weight loss and risk-factor management are known to improve the outcome of ablation, but lifestyle changes are often difficult to achieve in routine care.

Semaglutide (Wegovy®) is a GLP-1 receptor agonist approved in the EU for weight management. It has been shown to produce substantial and sustained weight loss and to improve metabolic and cardiovascular risk factors. Whether treatment with semaglutide before AF ablation can improve long-term rhythm outcomes has never been tested in a randomized clinical trial.

The WAIT-AF study is a randomized, open-label trial with blinded endpoint assessment. The study includes adults with AF who are scheduled for their first catheter ablation and have a BMI ≥30 kg/m², or ≥27 kg/m² with at least one additional cardiovascular risk factor (such as hypertension, diabetes and dyslipidemia). A total of 200 participants will be enrolled.

Participants are randomly assigned in a 1:1 ratio to either standard care or semaglutide (plus lifestyle advice) prior to their scheduled ablation. Semaglutide is administered according to the approved EU label with gradual dose escalation. All participants receive an implantable loop recorder (ILR) before ablation to continuously monitor heart rhythm throughout the study.

The primary objective is to determine whether semaglutide improves arrhythmia-free survival 12 months after AF ablation. Recurrence is defined as AF, atrial flutter, or atrial tachycardia lasting ≥30 seconds on continuous ILR monitoring, excluding the standard 3-month blanking period.

Secondary outcomes include weight loss, changes in blood pressure, AF symptoms, quality of life, AF burden, need for repeat ablation, hospitalizations for cardiovascular causes, and changes in metabolic risk factors. The study also evaluates safety and tolerability of semaglutide in this patient population.

The study aims to determine whether targeted weight management with semaglutide before AF ablation can improve long-term rhythm outcomes and overall cardiovascular health. If successful, this strategy may offer a new approach to optimizing treatment and improving the results of catheter ablation for patients with AF and overweight or obesity

DETAILED DESCRIPTION:
The WAIT trial evaluates whether metabolic optimization with once-weekly semaglutide prior to catheter ablation can improve rhythm outcomes in patients with atrial fibrillation and overweight/obesity. Excess adiposity and related cardiometabolic risk factors are strongly linked to atrial structural remodeling and higher rates of post-ablation arrhythmia recurrence. Although weight reduction is recommended in guidelines, sustained lifestyle-based weight loss is often difficult to achieve. Semaglutide provides an evidence-based pharmacologic strategy for clinically meaningful weight loss and risk-factor improvement, which may enhance the effectiveness of ablation.

This randomized, open-label study allocates participants 1:1 to semaglutide plus standard of care or standard of care alone for at least three months before undergoing their first AF ablation. All participants receive routine clinical management and continuous rhythm monitoring using an implantable loop recorder for 12 months post-ablation, with blinded adjudication of rhythm outcomes. The study integrates real-world clinical practice, using only routine clinical assessments, registry data, and ILR monitoring without introducing additional invasive procedures.

The trial is designed to determine whether targeted periablation metabolic therapy can increase arrhythmia-free survival, reduce AF burden, improve symptoms and quality of life, and favourably impact cardiovascular risk profiles. Results are expected to inform the role of GLP-1 receptor agonist therapy as part of a structured periablation optimization strategy for patients with AF and overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial, subjects must meet all of the following criteria:

1. Provision of written informed consent prior to participation.
2. Age ≥18 years.
3. Scheduled for first-time catheter ablation for atrial fibrillation using a pulmonary vein isolation (PVI) technique.
4. Body Mass Index (BMI) ≥30 kg/m² (obesity) OR

   BMI ≥27 kg/m² (overweight) with one or more of the following comorbidities:
   * prediabetes (defined as HbA1c 39-47 mmol/mol or fasting glucose 5,6-6,9 mmol/L),
   * known diabetes type 2
   * known hypertension (prior diagnosis and/or treatment with antihypertensive medication)
   * new diagnosis of hypertension (according to ESC GL for hypertension: Systolic BP ≥140 mmHg and/or diastolic BP ≥ 90 mmHg based on two readings on two separate visits, OR Ambulatory BP monitoring (24h average) ≥ 130/80 mmHg)
   * dyslipidemia defined as either one of the following

     * Known diagnosis of hyperlipidemia or
     * Treatment with lipid lowering medication

   OR either of the following:
   * LDL > 3.0 mmol/l
   * Total cholesterol > 5 mmol/l
   * Triglycerides > 1.7 mmol/l
   * HDL (< 1 mmol/l if male, < 1.2 mmol/l if female) AND/OR

     * atherosclerotic cardiovascular disease (prior myocardial infarction (MI), stroke, or peripheral arterial disease with claudication and ankle-brachial index <0.85, prior revascularization, or amputation)
     * obstructive sleep apnea.
5. For women of childbearing potential: Inclusion after a highly sensitive negative pregnancy test and agreement to use highly effective contraception during the study period (e.g., hormonal contraception, intrauterine device, or barrier method combined with spermicide).

Exclusion Criteria:

* Morbid obesity (BMI >40 kg/m²).
* Current use of GLP-1 receptor agonist therapy or dual agonist therapy within 6 months before screening.
* Current use of DPP-IV inhibitors.
* Diabetes type 1
* Known intolerance or contraindication to semaglutide.
* History of pancreatitis or recurrent hypoglycemia.
* Uncontrolled diabetic retinopathy
* Severe renal failure (estimated glomerular filtration rate [eGFR] <15 mL/min/1.73 m² or in dialysis)
* Severe hepatic failure (decompensated liver disease Child-Pugh class C)
* Severe cardiac failure (NYHA class IV)
* Life expectancy <12 months.
* Inability to self-administer the investigational medicinal product.
* Prior catheter ablation procedure for atrial fibrillation.
* Pregnancy, breastfeeding, or planned pregnancy during or within two months after the study period.
* Participation in another interventional clinical trial within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia-free survival at 12 months after catheter ablation, excluding the 3-month blanking period, with recurrence defined as any ILR-detected AF, atrial flutter, or atrial tachycardia ≥30 seconds. | 12 months post-ablation
  Arrhythmia-free survival at 12 months after catheter ablation, excluding the 3-month blanking period, with recurrence defined as any ILR-detected AF, atrial flutter, or atrial tachycardia ≥30 seconds.

SECONDARY OUTCOMES:
AF burden | At ablation and at 12 months post-ablation.
  trial fibrillation burden measured by continuous implantable loop recorder monitoring, expressed as the percentage of time in AF during predefined assessment windows. AF burden will be evaluated prior to the ablation procedure and again at 12 months post-ablation to compare the effect of the intervention versus standard of care.
Per protocol analysis of the primary outcome | 12 months post-ablation
  Assessment of arrhythmia-free survival at 12 months post-ablation in participants who completed the study without major protocol deviations. Recurrence is defined identically to the primary ITT analysis (ILR-detected AF, atrial flutter, or atrial tachycardia ≥30 seconds after the blanking period). This analysis evaluates the treatment effect under optimal adherence.
Time to first arrhythmia recurrence after the blanking period | From month 3 to month 12 post-ablation.
  Time from the end of the 3-month post-ablation blanking period to the first ILR-detected episode of atrial fibrillation, atrial flutter, or atrial tachycardia lasting ≥30 seconds. This endpoint evaluates the durability of rhythm control beyond the blanking period.
Number of repeat ablations required to achieve sinus rhythm | From index ablation to 12 months post-ablation.
  Total number of additional catheter ablation procedures performed per participant after the index ablation in order to restore or maintain sinus rhythm. This endpoint compares the need for redo ablations between the intervention and standard-of-care groups.
Freedom from symptomatic AF without redo ablation | From index ablation to 12 months post-ablation.
  Proportion of participants who remain free from symptomatic atrial fibrillation, atrial flutter, or atrial tachycardia without requiring a repeat ablation procedure. Symptomatic episodes are defined by patient-reported symptoms corroborated by rhythm documentation. This endpoint evaluates clinically meaningful rhythm control without the need for additional invasive therapy.
Symptom burden using questionnaires at baseline, ablation, 12 months | At baseline, at the time of ablation, and at 12 months post-ablation
  Assessment of atrial fibrillation-related symptom burden and functional impact using the AFEQT and AFSS validated questionnaires. Changes in symptom and quality-of-life scores will be compared between groups to evaluate improvement over time.
Quality of life changes using RAND-36 | At baseline, at the time of ablation, and at 12 months post-ablation.
  Assessment of changes in health-related quality of life using the RAND-36 questionnaire. .A clinically meaningful change is defined as an improvement of approximately 3-5 points in any RAND-36 domain. This endpoint evaluates the impact of the intervention on physical, emotional, and functional well-being over time.
Weight loss ≥10% or BMI <27 kg/m² at time of ablation and at 12 months post ablation | At the time of ablation and at 12 months post-ablation.
  Proportion of participants achieving either ≥10% reduction in baseline body weight or a BMI <27 kg/m². This endpoint assesses the metabolic effect of the intervention compared with standard of care.
Blood pressure reduction | At baseline, at the time of ablation, and at 12 months post-ablation.
  Change in systolic and diastolic blood pressure compared with baseline, including the proportion of participants achieving >10% systolic blood pressure reduction. Measurements are performed using standardized clinical procedures to evaluate the intervention's impact on blood pressure control.
Changes in blood biomarkers including glucose levels, HbA1c, creatinine and NT-proBNP | At routine clinical assessments nearest to baseline, ablation, and 12 months post-ablation.
  Evaluation of changes in fasting glucose and/or HbA1c and/or creatinine and/or NT-proBNP among participants with where these have been obtained through routine clinical care. This endpoint assesses whether the intervention influences glycaemic control and renal function l in patients for whom such measurements are already clinically indicated. No additional study-specific blood tests are performed.
Complications during and after the ablation procedure | During the ablation procedure and through 12 months post ablation.
  Incidence of procedure-related complications occurring during the catheter ablation or within the post-procedural follow-up period. Events may include vascular complications, pericardial effusion, tamponade, stroke/TIA, transient arrhythmias, anesthesia-related events, or other clinically relevant adverse outcomes, as documented in medical records. This endpoint compares procedural safety between study groups.
Left ventricular ejection fraction (LV-EF) pre- and post-ablation | At routine clinical echocardiography closest to baseline and the post-ablation assessment (up to 12 months).
  Assessment of changes in left ventricular ejection fraction from before to after the ablation procedure, based solely on echocardiograms performed as part of routine clinical care. No study-specific imaging is required; data will be included only for participants who undergo a post-ablation echocardiogram in standard practice. This endpoint evaluates whether the intervention influences cardiac function over time.
Prevalence of diabetes, renal failure, and heart failure | At baseline and at 12 months post-ablation (via clinical records and registry data).
  Assessment of the proportion of participants with diabetes, renal failure, or heart failure using information from routine clinical care, medical records, and linked registry data. No study-specific testing is performed. This endpoint describes baseline comorbidity burden and identifies new or worsening diagnoses captured through standard care or registries.
Cardiovascular hospitalization | From index ablation to 12 months post-ablation.
  Incidence of hospitalizations due to cardiovascular causes, identified through routine clinical records and national or regional registry data. Events may include admissions for arrhythmias, heart failure, acute coronary syndromes, or other cardiovascular conditions. No study-specific assessments are required.
All-cause hospitalization | From index ablation to 12 months post-ablation.
  Incidence of hospital admissions for any cause, identified through routine clinical records and national or regional registry data. This endpoint evaluates the broader healthcare impact of the intervention beyond cardiovascular events. No study-specific assessments are required.
Change in antiarrhythmic drug use | From baseline to 12 months post-ablation.
  Assessment of initiation, discontinuation, or dose changes in antiarrhythmic medications (e.g., class I or III agents, beta-blockers) based on routine clinical records. This endpoint evaluates differences in pharmacologic rhythm control requirements between groups.
Ablation procedure duration | During the index ablation procedure.
  Total duration of the catheter ablation procedure, extracted from routine procedural reports. This endpoint evaluates whether pre-ablation metabolic optimization influences procedural complexity.
Fluoroscopy time and radiation dose | During the index ablation procedure.
  Total fluoroscopy exposure time and radiation dose recorded during the index ablation procedure, as documented in routine procedural logs. This endpoint assesses potential differences in radiation exposure related to patient characteristics or weight loss.
Healthcare utilization | From randomization to 12 months post-ablation.
  Assessment of overall healthcare use, including outpatient cardiology visits, emergency department visits, and telephone/remote consultations. Data will be obtained from routine clinical records and linked regional or national healthcare registries. This endpoint evaluates whether the intervention affects healthcare demand and resource use. No study-specific visits or assessments are required.

OTHER OUTCOMES:
Artificial-intelligence based prediction of arrhythmia recurrence from 12-lead ECG | ECGs recorded as part of routine care at baseline, at ablation, and during follow-up up to 12 months post-ablation
  Exploratory assessment of whether artificial intelligence (AI) analysis of standard 12-lead ECGs can predict arrhythmia recurrence after ablation. ECGs obtained through routine clinical care will be analysed using validated AI algorithms to evaluate associations between ECG-derived features and later recurrence captured by ILR monitoring. No study-specific ECGs are required.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Svennberg, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to GDPR and national data protection regulations, the use of identifiable clinical and registry-linked data, and the absence of a fully anonymised IPD-sharing infrastructure. Data will only be accessible to authorised study personnel and regulatory bodies as required. Summary results will be published in accordance with scientific and ethical standards.